CLINICAL TRIAL: NCT06579924
Title: Re-usable Versus Disposable Rigid Nephroscope During Mini-PCNLs When Treating Large-burden Kidney Stones: an Feasibility Randomised Controlled Trial
Brief Title: Disposable Versus Disposable Nephroscope During PCNLs: a Feasibility RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DisposableRCTStudy
Record Dates: First submitted 2024-08-11; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Stone, Kidney
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mini-PCNL with disposable scope (Experimental): PCNLs carried out using disposable scope
  Interventions: Procedure: Disposable mini-PCNL
- Mini-PCNL using re-usable scope (Active Comparator): Mini-PCNLs carried out using re-usable scope
  Interventions: Procedure: Re-usable mini-PCNL

INTERVENTIONS:
Procedure: Disposable mini-PCNL — Mini-PCNL carried out using disposable scope
  Arms: Mini-PCNL with disposable scope
Procedure: Re-usable mini-PCNL — Mini-PCNL carried out using re-usable scope
  Arms: Mini-PCNL using re-usable scope

SUMMARY:
A feasibility randomised controlled trials comparing re-usable versus disposable nephroscope when treating kidney stones during mini-PCNLs

DETAILED DESCRIPTION:
Study Participants Patients undergoing minimally-invasive PCNLs with intention to treat renal low- to medium-burden renal stones.

Inclusion Criteria

* Patients undergoing mini PCNL to treat renal stones with a cumulative stone diameter 2-5 cm and completing at least a 3 month's follow-up
* Cases performed by surgeons beyond their learning curves
* Patients aged > 18
* Unenhanced CT scan carried out within 3 months pre-operatively
* Post-operative follow-up carried out according to our study protocol, with NCCT carried out within 2-3 months after surgery
* ASA 1-2
* Patients with normal weight (BMI: 18-25)
* Participant is willing and able to give informed consent to the proposed surgical treatment and agreeing to be enrolled in the study.

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

* Contraindications to surgical treatment
* PCNL performed for proximal ureteric stones
* Urinary tract with abnormal anatomy
* Obese patients
* ASA>3
* Patients with pyonephrosis
* Patients on anticoaugulants
* Preoperative CT scan not within 3 months before surgery
* Pregnant patients
* Patients younger than 18 years of age Study design and pathway The study will include patients with renal stones and undergoing mini-PCNL. All patients should respect inclusion/exclusion criteria. An ultra-low dose unenhanced CT scan (NCCT) has to be available for all cases pre-operatively, the post-operative follow-up will include NCCT within 2-3 months from treatment.

Patients will complete the study at 3 months post-op when the stone free rate will be assessed. Additionally, 30 days post-op complications will be recorded using Clavien-Dindo system. 3 months post-op stone-related events will be also registered.

Prior to enroll patients, participating surgeons will be asked to carry out 5 mini-PCNLs with disposable scope, aiming to render them more familiar and achieve learning curve.

Once the RCT will start, patient will be randomized in two groups using computer software (disposable group arm and non-disposable group arm).

Peri-operative data collection Peri-operative data will be collected using a standardized excel database produced by main investigator site.

The Stone complexity will be calculated according to database. Each case should be evaluated by two experienced surgeons and appropriate scoring should be agreed.

30 days post-operative complications should be recorded and reported using Clavien-Dindo classification System in its modified version for PCNLs. Type of complication in each Centre should be agreed by two different surgeons.

Post-operative patients' quality of life will be evaluated using validated version of WISQoL in Chinese7. It will be measured at 24 hours and 7 days post-op.

Definition of Stone free State: no > or equal to 2mm residual fragments (measured with post-operative NCCT). Size of residual fragments should be agreed with radiologist.

PCNL-Trifecta achievement will also be recorded.

Stone burden measurement

Authors will report maximum stone diameter and stone complexity reported using Guy's8 and S.T.O.N.E. nephrolithometry Score9. Stone characteristics should be agreed by two different surgeons. If multiple stones are present, the sum of their volume should be reported.

Surgical technique

Patients deemed suitable and enrolled in the study, will be operated as per routinary technique. This will include a prone position and placement of a retrograde 5-6 Fr ureteric catheter for pyelogram and dilatation of the urinary tract.

The puncture will be carried out according to surgeon's preference (under ultrasound, fluoroscopy or combination).

The track preparation will be carried out with one-shot dilator, if necessary progressive dilatation can be conducted. The percutaneous sheath will be 18 Fr.

The Single-Use Video Cystoscope RP-U-C0102 without bendable tip produced by (Redpine) will be used as rigid nephroscope in disposable group arm. This device has already obtained approval for endoluminal surgeries in China as well as CE and FDA approval for utilization in Western countries. In the non-disposable group, an equivalent size Hawk nephroscope will be used in the non-disposable arm.

The lithotripsy will be done with Ho-YAG laser, using a 550-micron laser fiber or ballistic lithotripter is believed appropriate.

In both arms, the percutaneous sheath will be 18 Fr peel-away sheath. Cases can be conducted tubeless or totally tubeless if necessary. If believed appropriate, in the group of patients treated with disposable cystoscope, surgeons are allowed to switch to a reusable nephroscope for any reason (which will be documented).

Definition of investigated complications

Complications will be categorized using Clavien-Dindo system. Authors will also specifically investigate bleeding and infective complications.

Infectious complications will include:

* Infection will be defined as temperature above 38C for a minimum of 24 hours and/or procalcitonin > 0,5 ng/mL and/or reactive C protein > 10.
* Septic shock: diagnosed using qSOFA Score
* ICU admission for sepsis
* Death
* Perirenal abscess

Hemorragic complications will include:

* Transfusion
* Hemoglobin drop >2 gr/dL
* Angioembolization
* Bleeding requiring secondary operation (bladder washout, ureteric stent positioning)
* Emergency nephrectomy for uncontrollable bleeding
* Hypovolemic shock requiring ICU stay

Study population

A total of 100 procedures will be included. The study will involve three surgeons. Each surgeon will carry out 20 procedures, 10 for each arm. The numerosity has been arbitrarily decided and in line with characteristics of pilot studies, aiming to test feasibility of disposable PCNLs and estimate numerosity for future RCT on this topic Before enrolling patients, all participating surgeons will be asked to carry out 5 mini-PCNLs with disposable scopes to render them familiar with the procedure and adjust the learning curve.

Statistical analysis The Statistical Package for the Social Sciences (SPSS) 20 will be used for statistical analysis.

Continuous variables will be presented as means (SDs) in cases of normal distribution and compared using the independent Student's t-test, while as median and interquartile range (IQR) in cases of skewed distributions and compared using the Mann-Whitney U-test. Categorical variables will be presented as numbers with percentages and compared using chi-square or Fisher's exact tests. Statistical significance will be considered for two-tailed P values of <0.05.

Endpoints As primary endpoints, authors will evaluate adequacy of disposable scopes (evaluating need to switch to re-usable scopes due to breakages, inadequacy, failures) and Stone Free Rates.

Authors will also collect as secondary endpoints complication rates and patients comfort, using WISQoL questionnaires.

Additionally, authors will use Likert scales to evaluate surgeons' appreciation (view, handling and weight of the instruments, irrigation, stability of the instrument, position and functionality of working channels).

Authors will also monitor the number procedures where there will be need of switching to re-usable scopes (due to malfunctioning/breakage/inadequacy of disposable scopes).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mini PCNL to treat renal stones with a cumulative stone diameter 2-5 cm and completing at least a 3 month's follow-up
* Cases performed by surgeons beyond their learning curves
* Patients aged > 18
* Unenhanced CT scan carried out within 3 months pre-operatively
* Post-operative follow-up carried out according to our study protocol, with NCCT carried out within 2-3 months after surgery
* ASA 1-2
* Patients with normal weight (BMI: 18-25)
* Participant is willing and able to give informed consent to the proposed surgical treatment and agreeing to be enrolled in the study.

Exclusion Criteria:• Contraindications to surgical treatment

* PCNL performed for proximal ureteric stones
* Urinary tract with abnormal anatomy
* Obese patients
* ASA>3
* Patients with pyonephrosis
* Patients on anticoaugulants
* Preoperative CT scan not within 3 months before surgery
* Pregnant patients
* Patients younger than 18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 90 days post-op
  ability of used scope in determining a complete stone clearance, or absence of clinically significant residual fragments

SECONDARY OUTCOMES:
complication rate | 30 days post-op
  presence of post-operative complications according to Calvin-Dindo classification system
adequacy of used instrument | intra-operative assessment
  adequacy of instruments (including failure, quality of view, handling) will be tested

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No